CLINICAL TRIAL: NCT04127630
Title: Evaluation in MRI of the Impact of the Sellick Manoeuvre or Para-tracheal Compression of the Cervical Esophagus on the Displacement of the Laryngeal Mass and the Visualization of the Vocal Cords
Brief Title: MRI STUDY OF THE LPEC
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Other Study IDs: ANESAM2019
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mobilization of the larynx: we aim to asses with an magnetic resonance imaging the compressibility of the oesophagus with LPEC
  Interventions: Procedure: mobilization of the larynx

INTERVENTIONS:
Procedure: mobilization of the larynx — we aim to asses with an magnetic resonance imaging the compressibility of the oesophagus with LPEC

SUMMARY:
Cricoid pressure is still considered as a standard of care in order to prevent the gastric regurgitation in full stomach surgery1.

However, this attitude has been challenged in several case reports as oesophageal rupture, difficult intubation, and even failing to occlude the oesophagus. Moreover, in a large prospective randomized study , this maneuver has failed to show a definite benefit2.

The lateral deviation to the left of the oeso deviate to the left side3,4 has led to the description of a new maneuver to compress directly the oesophagus at the low left paratracheal level. This maneuver has been shown to prevent gastric air insuflation during the ventilation.

In the present study, the investigators aim to asses with an magnetic resonance imaging the compressibility of the oesophagus.

ELIGIBILITY:
Inclusion Criteria:

* Adults Volunteers

Exclusion Criteria:

* Pregnancy
* Claustrophob
* Thyroid goiter

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Oesophagus compressibility | End of the MRI
  Analysis of the position of the Oesophagus is obtained in the three groups in a upper position ( C5-6) and lower position (C8-T1). The upper position is the first view were the oesophagus is clearly identified: In fact, the pressure exerted during the cricoid maneuver is in fact applied in the area of the hypopharynx above the osophagus. The oesophagus is quoted relatively to the vertebral body as Medial (80% facing the vertebral body) Medio-lateral , lateral (20% facing the vertebral body).

CONTACTS AND LOCATIONS:
Locations (1):
- Javillier, Liège, Belgium